CLINICAL TRIAL: NCT06070597
Title: Effects of Iclepertin on the QT Interval Following Oral Administration in Healthy Male and Female Subjects (a Double-blind, Randomised, Placebo-controlled, Multiple-dose, Parallel Group With Nested Crossover Design Trial, With Moxifloxacin as Positive Control)
Brief Title: A Study in Healthy People to Test Whether Iclepertin Has an Effect on Cardiac Safety
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1346-0051; 2023-504693-38-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: A double-blind, randomised, placebo-controlled, multiple-dose, parallel group with nested crossover design trial, with moxifloxacin as positive control
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Iclepertin treatment+ Placebo to Moxifloxacin (Experimental): Placebo to moxifloxacin (Day 1) + Iclepertin (Day 1-12) + Placebo to moxifloxacin (Day 13
  Interventions: Drug: Iclepertin; Drug: Moxifloxacin Placebo
- Arm B1: Iclepertin Placebo treatment + Moxifloxacin (Experimental): Moxifloxacin (Day 1) + Placebo to iclepertin (Day 1-12) + Placebo to moxifloxacin (Day 13) - Arm B1
  Interventions: Drug: Iclepertin Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo
- Arm B2: Iclepertin Placebo treatment + Placebo to Moxifloxacin (Experimental): Placebo to moxifloxacin (Day 1) + Placebo to iclepertin (Day 1-12) + Moxifloxacin (Day 13) - Arm B2
  Interventions: Drug: Iclepertin Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Placebo

INTERVENTIONS:
Drug: Iclepertin — Iclepertin
  Arms: Arm 1: Iclepertin treatment+ Placebo to Moxifloxacin
Drug: Iclepertin Placebo — Placebo to Iclepertin
  Arms: Arm B1: Iclepertin Placebo treatment + Moxifloxacin; Arm B2: Iclepertin Placebo treatment + Placebo to Moxifloxacin
Drug: Moxifloxacin — Moxifloxacin
  Arms: Arm B1: Iclepertin Placebo treatment + Moxifloxacin; Arm B2: Iclepertin Placebo treatment + Placebo to Moxifloxacin
Drug: Moxifloxacin Placebo — Placebo Moxifloxacin

SUMMARY:
This study aims to evaluate the effects of iclepertin in the range of therapeutic to supra-therapeutic exposures on the (QT/QTc): Electrocardiogram (ECG) time interval from the start of the QRS complex (ECG time interval) to the end of the T wave / QT interval corrected for heart rate, e.g. using the method of Fridericia or Bazett interval and other ECG parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, ital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests without clinically significant abnormalities
2. Age of 18 to 50 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
5. Either male subject, or female subject who meets any of the following criteria for a highly effective contraception from at least 30 days before the first administration of trial medication until 30 days after trial completion:

   * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal, subdermal or transdermal), plus condom
   * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants), plus condom
   * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
   * Sexually abstinent
   * A vasectomized sexual partner who received medical assessment of the surgical success (documented absence of sperm) and provided that partner is the sole sexual partner of the trial participant
   * Surgically sterilized (including hysterectomy)
   * Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of Follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L (or the reference range from the local safety laboratory) is confirmatory), hormone replacement therapy is not permitted Note: Male subjects are not required to use contraception.

Exclusion Criteria:

Subjects will not be allowed to participate, if any of the following general criteria apply:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance, in particular, hepatic parameters (Alanine transaminase (ALT), Aspartate aminotransferase (AST), total bilirubin) or renal parameters (creatinine) exceeding the Upper limit of normal (ULN)
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts

Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
QTcF change from baseline matched to the plasma concentration of iclepertin collected at the same time point | Up to 12 days
  QT interval corrected for heart rate, e.g. using the method of Fridericia (QTcF).

SECONDARY OUTCOMES:
QTcF change from baseline matched to the plasma concentration of moxifloxacin collected at the same time point | Up to 1 day
  QT interval corrected for heart rate, e.g. using the method of Fridericia (QTcF).

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com